CLINICAL TRIAL: NCT00538356
Title: IN-TIME: Influence of Home Monitoring on the Clinical Status of Heart Failure Patients
Brief Title: Influence of Home Monitoring on the Clinical Status of Heart Failure Patients With an Impaired Left Ventricular Function
Acronym: IN-TIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS042; There is no secondary ID
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia; Congestive Heart Failure
Keywords: Heart failure; Rehospitalization:; Packer composite score; Home Monitoring; Cardiac resynchronization therapy; Implantable cardioverter-defibrillator
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular; Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Monitoring (Experimental): ICD or CRT-D with Home Monitoring feature activated Home Monitoring data will be analyzed regularly and patients will be contacted and scheduled for additional follow-up after predefined events
  Interventions: Device: ICD or CRT-D with Home Monitoring feature activated
- Control (Active Comparator): ICD or CRT-D with Home Monitoring feature deactivated Patients will be treated as per standard of care in each participating clinic
  Interventions: Device: ICD or CRT-D with Home Monitoring feature deactivated

INTERVENTIONS:
Device: ICD or CRT-D with Home Monitoring feature deactivated — Standard care
  Arms: Control
Device: ICD or CRT-D with Home Monitoring feature activated — Standard care + patient management by Home Monitoring
  Other Names: Biotronik Home Monitoring; Home Monitoring Service Center
  Arms: Home Monitoring

SUMMARY:
Re-hospitalizations or deaths by worsening heart failure are often preceded by distinct trends of clinical parameters such as atrial or ventricular arrhythmia, activity, heart rate variability, or ventricular ectopy. The Home Monitoring™ capability offered by BIOTRONIK active implants has the potential to detect some of these trends early and thus to offer the possibility to intervene in time for prevention of fatal worsening of heart failure.

To investigate the predictive value of Home Monitoring parameters, patients with symptomatic heart failure and reduced ejection fraction receiving an implantable cardioverter-defibrillator (ICD) or an ICD in combination with cardiac resynchronization therapy (CRT-D) will be randomized between prospective patient management by Home Monitoring analysis or standard care. The influence of Home Monitoring on the clinical status of heart failure patients will be assessed.

DETAILED DESCRIPTION:
Hospital admissions or deaths by worsening heart failure are often preceded by distinct trends of clinical parameters such as heart rhythm disturbances, daily physical activity of a patient, or mean heart rates.

The Home Monitoring™ capability offered by many BIOTRONIK implants has the potential to detect some of these trends early. During Home Monitoring surveillance, medical and technical data from an ICD or CRT device are sent to a modified mobile phone, the so-called Cardio Messenger. This device transmits the data via a mobile phone network to the BIOTRONIK service center. There, the data are put into an easily accessible form and can then be viewed by the physician online via the internet on a secure website. Additionally, the occurrence of heart rhythm disturbances or device problems will be transmitted by fax, SMS or email.

This unique system allows the attending physician to monitor each patient very closely and to react early enough to prevent worsening of heart failure at an early stage, to optimize therapy, and to secure the correct functioning of the implant.

The goal of IN-TIME is thus to analyze the impact of a regular Home Monitoring evaluation on the health status of heart failure patients receiving such an implant as part of their therapy.

A total of 720 patients with heart failure symptoms and a severely reduced pumping function receiving an ICD or a CRT-D device from up to 50 European clinical centers will be enrolled into the study. About 4 weeks after discharge from the implanting hospital, patients will be randomly assigned to prospective patient management by Home Monitoring or standard care groups. Patients in the Home Monitoring group will be monitored at least once per week, patients in the control group will not be monitored during the study, but their transmitted Home Monitoring data will be analyzed after their ending of participation in the study.

The health status of patients will be measured using the well established "Packer Score". This score is a combined measurement of death rates, hospital admission rates, heart failure symptom classification and quality of life. Patients will be classified at their end of study participation as worsened, unchanged, or improved based on these parameters. To this end, the health status of participating patients will be determined regularly during further outpatient follow ups. These will take place at regular intervals due to the standard care.

Additionally, some special parameters sent to the physician via Home Monitoring will be analyzed whether they could possibly predict an imminent worsening of a patient's health - leading to an unplanned hospital visit - so that it could perhaps be prevented in the future.

Patients remain within the study for 12 months after randomization or until their participation is ended prematurely, e.g. by withdrawal of their consent, a low data transmission rate, or death.

ELIGIBILITY:
Inclusion Criteria:

* Indication for single chamber ICD, dual chamber ICD or CRT-D
* Chronic heart failure (≥ 3 months)
* NYHA Class II or III for 1 month prior to screening
* LVEF ≤ 35% within 3 months prior to screening
* Indication for therapy with diuretics
* Patient informed consent

Exclusion Criteria:

* Uncontrolled hypertension
* NYHA class I or IV
* Permanent atrial fibrillation
* Life expectancy < 1 year
* Restrictive, infiltrative or hypertrophic cardiomyopathy, constrictive pericarditis, acute myocarditis
* Severe mitral regurgitation
* Symptomatic aortic stenosis
* Tricuspid valve replacement
* Known drug or alcohol abuse
* Expected non-compliance
* Pregnancy
* Participation in another telemonitoring concept
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2007-07; Primary Completion 2012-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Composite Score of death, hospitalization for heart failure, NYHA class and global assessment (Packer Score) | 12 months

SECONDARY OUTCOMES:
Rehospitalizations due to worsening heart failure; Correlation of Home Monitoring values with the clinical status; Incidence and reasons for Home Monitoring based interventions; Home Monitoring workflow analysis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Prof. Dr., Study Chair — Herzzentrum Leipzig, Germany
Locations (39):
- Sydney Adventist Hospital, Wahroonga, Australia
- Universitätsklinik für Innere Medizin, Innsbruck, Austria
- Czechia (2):
  - Institute of Clinical and Experimental Medicine, Prague
  - Hospital Na Homolce, Prague
- Denmark (4):
  - Aalborg Hospital, Aalborg
  - Århus Universitetshospital, Skejby Sygehus, Århus N
  - Gentofte Hospital, Hellerup
  - Odense Universitets Hospital, Odense
- Germany (27):
  - Zentralklinik Bad Berka, Bad Berka
  - Herz- und Gefäßklinikum Bad Neustadt GmbH, Bad Neustadt an der Saale
  - Bad Segeberger Kliniken GmbH, Bad Segeberg
  - Vivantes Klinikum Neukölln, Berlin
  - Vivantes Klinikum am Urban, Berlin
  - Universitätsklinikum Charité Campus Benjamin Franklin, Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - Städtische Kliniken Bielefeld, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Coburg gGmbH, Coburg
  - Klinikum Lippe-Detmold, Detmold
  - Westdeutsches Herzzentrum des Universitätsklinikums Essen, Essen
  - Universitätsklinikum Gießen und Marburg, Giessen
  - Medizinische Hochschule, Hanover
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Klinikum St. Georg gGmbH, Leipzig
  - Herzzentrum der Universität Leipzig, Leipzig
  - Universitätsklinik Schleswig-Holstein, Lübeck
  - St. Marienhospital Lünen GmbH, Lünen
  - Klinikum Schwabing, Kardiologie, Munich - Schwabing
  - Kardiologische Gemeinschaftspraxis Dr. Mühling, München
  - Stiftsklinik Augustinum, Innere Medizin / Kardiologie, München
  - Klinikum der Universität München Großhadern, München
  - Herzzentrum München-Bogenhausen, München
  - Kardiologische Gemeinschaftspraxis Dr. Predel, Dr. Heinrich, Nordhausen
  - St. Vincenz Krankenhaus GmbH, Paderborn
  - Klinikum Pirna GmbH, Pirna
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Tel Litwinsky
- P. Stradins Clinical University Hospital, Latvian Centre of Cardiology, Riga, Latvia

REFERENCES:
- [Background] Arya A, Block M, Kautzner J, Lewalter T, Mortel H, Sack S, Schumacher B, Sogaard P, Taborsky M, Husser D, Hindricks G; IN-TIME investigators. Influence of Home Monitoring on the clinical status of heart failure patients: Design and rationale of the IN-TIME study. Eur J Heart Fail. 2008 Nov;10(11):1143-8. doi: 10.1016/j.ejheart.2008.08.004. Epub 2008 Sep 19. PMID 18805053
- [Derived] Hindricks G, Taborsky M, Glikson M, Heinrich U, Schumacher B, Katz A, Brachmann J, Lewalter T, Goette A, Block M, Kautzner J, Sack S, Husser D, Piorkowski C, Sogaard P; IN-TIME study group*. Implant-based multiparameter telemonitoring of patients with heart failure (IN-TIME): a randomised controlled trial. Lancet. 2014 Aug 16;384(9943):583-590. doi: 10.1016/S0140-6736(14)61176-4. PMID 25131977